CLINICAL TRIAL: NCT05285098
Title: Retrospective Analysis of 15 Years of Leipzig "Fast-Track" Concept.
Brief Title: Leipzig FAST-TRACK Over 15 Years for Cardiac Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FT15
Record Dates: First submitted 2022-01-31; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Post-cardiac Surgery
Keywords: Fast track after cardiac surgery; ERAS cardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since November 2005, we are running a specialized post anesthetic care unit (PACU) in our tertiary, university affiliated high-volume heart centre. In our concept, we are bypassing ICU admission completely. The fast-track concept was initially applied to pre-selected elective patients undergoing low-risk operations. However, promising outcomes led to a more widespread utilization with more complex procedures. The aim of this study is to analyse the fast track evolutions.

DETAILED DESCRIPTION:
Fast Track Treatment includes many elements recommended by the ERAS Society for cardiac surgery(1). Since November 2005, we are running a specialized post anesthetic care unit (PACU) in our tertiary, university affiliated high-volume heart centre. In our concept, we are bypassing ICU admission completely. The patients are transferred from the operation room to the recovery room, extubated there within a short time, stabilized and transferred on the same day to intermediate care (IMC). Ideally, the patient will be transferred to the normal ward on the first postoperative day. The fast-track concept was initially applied to pre-selected elective patients undergoing low-risk operations. However, promising outcomes led to a more widespread utilization with more complex procedures. The aim of this study is to analyse the evolutions within the fast-track protocol over a period of 15 years (from November 2005 to December 2020).

ELIGIBILITY:
Inclusion Criteria:

* Adults >18y

Exclusion Criteria:

* Incomplete data
* Catheter-valve implantation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: -All consecutive cardiac surgical patients treatet with Leipzig fast-track protocol
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
FT evolution analysis in complexity | Novmber 2005- December 2020
  Trends analysis in complexity ( using EUROSCORE II) against time (in years)
FT evolution analysis in length of stay | Novmber 2005- December 2020
  Trends analysis of length of stay ( in hospital and ICU in days) against time (in years)
FT evolution analysis in postoperative complications | Novmber 2005- December 2020
  Trends analysis in postoperative complications ( cardiac, pulmonary, and neurological) in percentage against time ( in years)
FT evolution analysis in postoperative mortality rate | Novmber 2005- December 2020
  Trends analysis of postoperative mortality rate ( in percentage) against time (in years)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Ender, Study Chair — Leipzig Heart center
Locations (1):
- Leipzig Heart center, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Retrospective analysis of the data ( collected from the hospital clinical information systems) for all consecutive patients admitted to PACU during 15 years.

REFERENCES:
- [Background] Ender J, Borger MA, Scholz M, Funkat AK, Anwar N, Sommer M, Mohr FW, Fassl J. Cardiac surgery fast-track treatment in a postanesthetic care unit: six-month results of the Leipzig fast-track concept. Anesthesiology. 2008 Jul;109(1):61-6. doi: 10.1097/ALN.0b013e31817881b3. PMID 18580173
- [Background] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Background] Wong WT, Lai VK, Chee YE, Lee A. Fast-track cardiac care for adult cardiac surgical patients. Cochrane Database Syst Rev. 2016 Sep 12;9(9):CD003587. doi: 10.1002/14651858.CD003587.pub3. PMID 27616189